CLINICAL TRIAL: NCT01535794
Title: Exploring the Potential for Social Network Site-delivered Interventions to Increase HPV Vaccine Uptake Among Men Who Have Sex With Men
Brief Title: HPV Vaccine Acceptability Among Young Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: YMSM HPV vaccine acceptability
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: HPV Vaccine Attitudes; HPV Vaccine Intention
Keywords: HPV vaccine; acceptability; males; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 18-26 year old men who have sex with men

SUMMARY:
The FDA has recently approved Gardasil for the prevention of anal cancer in people aged 9-26. Men who have sex with men (MSM) have disproportionately high rates of anal cancer and could benefit greatly from vaccination. Vaccine uptake among young MSM (YMSM) is poor, and little is known about factors associated with vaccine acceptance in this population. With the risk of anal cancer among MSM higher than the risk of cervical cancer among women before routine cytological screening was introduced, acceptance of a prophylactic vaccine in this subgroup is the most cost-effective and attainable strategy to greatly reduce the prevalence of anal cancer. While the investigators can assume the human papillomavirus (HPV) vaccine has many acceptable concepts among these men, there are multiple barriers which may potentially interfere with their likelihood of initiating the vaccine series. Vaccine catch-up rates among women of a similar age has been poor, and there is no reason to expect this to be higher among men. One potential strategy to increase vaccine uptake in this catch-up group is to implement a patient-driven program to promote vaccination among men.

This project will contribute to the investigators understanding of how the investigators can utilize social networks to identify barriers to HPV vaccination among YMSM, and how to potentially influence a patient-driven vaccination effort to increase uptake among men in the catch-up age group. This research will inform future interventions to targeted populations that may be incorporated into online social networking websites to encourage HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 18-26 years old
* male

Exclusion Criteria:

* younger than 18 years old
* older than 26 years old
* female

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be an internet-based, cross-sectional study targeting all US profiles of two separate online social/sexual networking communities of YMSM. A recruitment email will be sent internally to all active US profiles for men 18-26 years old.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
HPV vaccine acceptability | Spring 2012
  The primary outcome in this study is young men's intention to be vaccinated for human papillomavirus (HPV). This will be measured on a scale of 0-100, with a higher number indicating greater likelihood of future vaccination. No vaccine will be administered.

SECONDARY OUTCOMES:
Attitudes towards HPV vaccination | Spring 2012
  A secondary outcome will be young men's attitudes towards HPV vaccination, including their beliefs about vaccine safety, efficacy, and effectiveness. This outcome will also assess the presence of logistical or pragmatic barriers to their future vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States